CLINICAL TRIAL: NCT01308905
Title: Pilot Study to Determine the Utility of [18F] 3&Apos;-Deoxy-3&Apos;-Fluorothymidine- Positron Emission Tomography in Monitoring Patient Response to Chemotherapy in Neuroblastoma
Brief Title: Monitor Response to Treatment in Neuroblastoma Using 3&Apos;-Deoxy-3&Apos;-Fluorothymidine- Positron Emission Tomography (FLT-PET)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: Children's Hospital of Michigan (Other)
Responsible Party: Principal Investigator, Zhihong Wang, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WSU 2009-031
Record Dates: First submitted 2011-02-22; First posted 2011-03-04 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Intervention Model Description: PET scans will be performed to show the distribution throughout the body of substances containing a small amount of radioactive material.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FLT-PET (Experimental): Patients will be managed per COG protocol ANBL00B1 (low risk, LR), ANBL0521 (intermediate risk, IR), ANBL0531 (high risk, HR) or other future neuroblastoma studies according to their risk group (risk assignment, treatment schema and protocols are available in COG website). The following is a brief description of the treatment.
  1. Low risk patients: observation only.
  2. Intermediate risk patients: chemotherapy stratified according to risk sub-groups followed by surgical resection.
  3. High risk patients: 6 courses of induction chemotherapy, surgical resection and high dose chemotherapy with autologous stem cell transplant (SCT), involved field radiation and 6 months of Isotrenitoin.
  PET scan will be conducted at diagnosis, at the end of the first cycle of treatment and prior to the surgical procedure (resection).
  Interventions: Device: FLT-PET

INTERVENTIONS:
Device: FLT-PET — PET scan will be conducted at diagnosis, at the end of the first cycle of treatment and prior to the surgical procedure (resection).

SUMMARY:
The purpose of this study is to gain knowledge about how to best diagnose and treat tumors, how tumors affect normal tissue and how treatment of tumors with radiation therapy and chemotherapy affect tumors.

DETAILED DESCRIPTION:
The purpose of this research study is to observe the changes within the tumor cells which may improve the understanding of how tumors grow and how they respond to various treatments. These changes will be compared with results of the physical examination and scans (CT and MRI) that are done as part of clinical care. Images will be made showing the distribution throughout the body of substances containing a small amount of radioactive material. This procedure is called a PET scan. The radioactive substances (tracer compound) in this study are [F-18] FLT.

ELIGIBILITY:
Inclusion Criteria:

* All patients with neuroblastoma or suspected neuroblastoma seen at Children's Hospital of Michigan (CHM). Patients need to be 2 years or older to be eligible for the initial study
* Patients must be 1 day to 21 years old, there is no gender limit.
* Diagnosis: All patients with neuroblastoma or suspected neuroblastoma, including newly diagnosed and relapsed patients, are eligible for Objective 1. To be eligible for Objective 2, patients must have a diagnosis of neuroblastoma verified by histology or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites, and have measurable disease after the initial surgery
* Female adolescent patients must have a negative pregnancy test within 14 days of first imaging and should not be pregnant
* Patients must be able to lie still for the tests, or have no contraindication for sedation
* Patients or their legal guardian must sign an informed consent indicating that they are aware of the investigational nature of this study
* A total number of 40-50 patients will be included in the study

Exclusion Criteria:

* Patients who do not have a histology diagnosis of neuroblastoma are not eligible for the study
* Patients whose definite diagnosis after surgery is not consistent with the diagnosis of neuroblastoma will be included in the Objective 1 but excluded for Objective 2.

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
To determine whether 18F-FLT-PET is a sensitive tool to image neuroblastoma. | 1st PET - At diagnosis

SECONDARY OUTCOMES:
To evaluate the utility of FLT-PET in early assessment of patient response to treatment. | 1st PET - At diagnosis
To evaluate the utility of FLT-PET in early assessment of patient response to | 2nd PET - Approx. 3 wks (end of 1st cycle)
To evaluate the utility of FLT-PET in early assessment of patient response to treatment. | 3rd PET: 6-15 wks (Prior to surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F. Shields, M.D., Ph.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States